CLINICAL TRIAL: NCT02310152
Title: Explanatory Clinical Trial of a Novel Parent Intervention for Childhood Anxiety (SPACE)
Acronym: SPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1311013020; 5K23MH103555-03 (NIH)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Anxiety Disorders; Anxiety, Separation; Phobic Disorders
Keywords: Child; Adolescent; Parents; Cognitive Therapy; Cognitive Behavior Therapy; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Anxiety, Separation; Phobic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment: CBT (Active Comparator): Cognitive Behavioral Therapy
  Interventions: Behavioral: CBT
- Experimental Treatment: SPACE (Experimental): Parent-Based Treatment of Childhood and Adolescent Anxiety Disorders
  Interventions: Behavioral: Parent-Based Treatment of Child and Adolescent Anxiety Disorders

INTERVENTIONS:
Behavioral: Parent-Based Treatment of Child and Adolescent Anxiety Disorders — Supportive Parenting for Anxious Childhood Emotions
  Other Names: SPACE
  Arms: Experimental Treatment: SPACE
Behavioral: CBT — Cognitive Behavioral Therapy
  Arms: Active Treatment: CBT

SUMMARY:
Childhood anxiety disorders are very common, carry tremendous personal and societal costs, frequently do not respond adequately to treatment, and involving parents in treatment has so far not enhanced outcomes. Explanatory clinical trials are needed to identify parent specific mechanisms of change that are not targeted in direct child treatment, and to identify markers of who is most likely to benefit from parent intervention. This study is an explanatory clinical trial of a parent based intervention and of cognitive behavioral therapy, and an investigation of biological and behavioral moderators of treatment response.

DETAILED DESCRIPTION:
Despite strong evidence for the efficacy of individual cognitive-behavior therapy (ICBT) for childhood anxiety disorders, up to 50% of children remain symptomatic after treatment and many still meet diagnostic criteria. Evidence for parental influences in the etiology and maintenance of anxiety in children has often led to the reasonable assumption that adding parent work to ICBT would enhance treatment effects. This idea has now been repeatedly tested in randomized controlled trials (RCTs) that compared ICBT to ICBT with added parent work. The specific content of the parent work has varied but has mainly included teaching parents skills for contingency management, modeling appropriate behavior, and reducing family conflict. Working with parents in these ways has so far not led to enhanced treatment effects compared to ICBT alone, as a number of meta-analytic and comprehensive reviews have shown.

One plausible conclusion from these data is that parent work cannot enhance effects beyond what is achieved through ICBT alone. This study focuses on an alternative plausible conclusion: That parent interventions need to be informed by theoretical working models of parent-specific mechanisms of change that are not targeted in ICBT; and that parent interventions need to be evaluated in explanatory RCTs that ask not only 'does treatment work?' but also 'how and for whom does treatment work?' Underlying systems that shape how parents respond to child anxiety or distress can provide clues to parent-specific targets for intervention and can point to potential moderators of treatment response. Identifying mechanisms by which parent interventions can enhance child anxiety outcomes, and identifying markers of parents most in need of such interventions advances the goal of personalized psychotherapy, and is the overall goal of this study.

Family accommodation (FA) describes parents' attempts to help a child avoid feeling anxious by participating in symptom-driven behaviors and modifying family routines. FA is highly prevalent among parents of anxious children and has been linked to greater symptom severity in the child and to poorer response to ICBT. Research has linked a number of biological and behavioral parent markers to protective parental behavior and to child anxiety. The nonapeptide oxytocin (OT) is implicated in parental attachment and protective behavior in humans and animals. Coded behavioral observations link aspects of parental behavior (i.e., autonomy granting, over involvement, and sensitivity) to child anxiety. A number of studies also have shown that these biological and behavioral markers interact to predict anxiety outcomes in at-risk children. Yet so far this research has been siloed from intervention research and has not informed parent-based treatments, highlighting the need for clinical investigators equipped with the necessary skills to integrate multiple units of analysis into explanatory RCTs of novel interventions.

This study represents a fusion of clinical, biological and behavioral research through an explanatory RCT of a parent-based treatment focused on modifying parental responses to child anxiety and distress as a mediator of treatment outcome, and on biological and behavioral markers as possible moderators of treatment outcome. The intervention evaluated in this study (Supportive Parenting for Anxious Childhood Emotions; SPACE) aims to systematically reduce FA through a series of concrete manualized steps. This study is an integrated explanatory RCT of SPACE with the following 3 specific aims:

Aim 1 - Specificity: Does SPACE lead to significantly lower levels of FA compared to ICBT? Hypothesis: Levels of FA for parents in SPACE will be significantly lower after treatment than before treatment, as compared to parents of children in ICBT.

Aim 2 - Mediation: Does reducing FA lead to positive child outcomes? Hypothesis: Parents' reduced FA will be a significant mediator of positive child outcomes (i.e., reduced child anxiety).

Aim 3 - Moderation: Do key biological and behavioral markers (i.e., parental OT, autonomy granting, over involvement, sensitivity) moderate child outcomes? Hypothesis: Baseline levels of maternal OT, autonomy granting, over involvement, and sensitivity will be significant moderators of child outcomes (i.e., reducing child anxiety).

ELIGIBILITY:
Inclusion Criteria:

Children:

* meet criteria for a primary DSM5 anxiety disorder of generalized anxiety disorder (GAD), social phobia (SOP), and separation anxiety disorder (SAD) using the DSM-5 version of the Anxiety Disorders Interview Schedule -Child and Parent Versions (ADIS-C/P)
* mean score of 4 or greater on the ADIS-C/P Clinician Rating Scale of Severity (CSR)
* ceasing all other psychosocial treatment upon consultation with the clinic staff and the service provider
* not using any psychotropic medication other than a stable dose of stimulant medication treatment for comorbid ADHD or a stable dose of Selective Serotonin Reuptake Inhibitor (SSRI)
* children who are on a stable dose of stimulant medication or SSRI (i.e., a minimum of six weeks at the same dose) will be included so as not to limit generalizability.

Exclusion Criteria:

Children:

* primary diagnosis of any Axis I DSM-IV disorder other than GAD, SOP, Phobias and SAD
* any of the following disorders (e.g., primary, secondary, tertiary) - Pervasive Developmental Disorders, Mental Retardation, Organic Mental Disorders, Bipolar Disorder, Schizophrenia and Other Psychotic Disorders
* drug or alcohol abuse/dependence will also be exclusionary
* tic disorders will not be exclusionary unless they require psychotropic medication to stabilize
* Significant active suicidal ideation or a past suicide attempt in the last 6 months. Adolescents with a history of non-lethal self-harm behaviors (e.g., cutting) will be allowed to enroll if they meet other criteria
* have an intellectual disability as reported by guardian
* be a victim of past or present undisclosed abuse requiring investigation or ongoing supervision by the Department of Social Services
* not have been cohabiting with mother for at least one year prior to admittance. Parent:
* any of the following disorders (e.g., primary, secondary, tertiary) - Pervasive Developmental Disorders, Mental Retardation, Selective Mutism, Organic Mental Disorders, Bipolar Disorder, Schizophrenia and Other Psychotic Disorders. Drug or alcohol abuse/dependence will also be exclusionary
* not have been cohabiting with child for at least one year prior to admittance
* report the presence of any active suicidal ideation or a past suicide attempt in the last 6 months.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2014-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scale Improvement and Severity | After 12 weeks of treatment
  Clinician determined rating of illness
Pediatric Anxiety Rating Scale | After 12 weeks of treatment
  Clinician administered rating of child anxiety

SECONDARY OUTCOMES:
Screen for Childhood Anxiety Related Disorders | After 12 weeks of treatment
  A self and parent report of child anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Lebowitz, E. R., Omer, H., Hermes, H., & Scahill, L. (2013). Parent Training for Childhood Anxiety Disorders: The SPACE Program. Cognitive and Behavioral Practice.
- [Background] Lebowitz ER, Woolston J, Bar-Haim Y, Calvocoressi L, Dauser C, Warnick E, Scahill L, Chakir AR, Shechner T, Hermes H, Vitulano LA, King RA, Leckman JF. Family accommodation in pediatric anxiety disorders. Depress Anxiety. 2013 Jan;30(1):47-54. doi: 10.1002/da.21998. Epub 2012 Sep 10. PMID 22965863
- [Derived] Lebowitz ER, Marin C, Martino A, Shimshoni Y, Silverman WK. Parent-Based Treatment as Efficacious as Cognitive-Behavioral Therapy for Childhood Anxiety: A Randomized Noninferiority Study of Supportive Parenting for Anxious Childhood Emotions. J Am Acad Child Adolesc Psychiatry. 2020 Mar;59(3):362-372. doi: 10.1016/j.jaac.2019.02.014. Epub 2019 Mar 7. PMID 30851397